CLINICAL TRIAL: NCT00689221
Title: Cilengitide for Subjects With Newly Diagnosed Glioblastoma and Methylated MGMT Gene Promoter - A Multicenter, Open-label, Controlled Phase III Study, Testing Cilengitide in Combination With Standard Treatment (Temozolomide With Concomitant Radiation Therapy, Followed by Temozolomide Maintenance Therapy) Versus Standard Treatment Alone (CENTRIC)
Brief Title: Cilengitide, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma and Methylated Gene Promoter Status
Acronym: CENTRIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 121974-011; EORTC 26071-22072; 2007-004344-78 (EudraCT Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Glioblastoma
Keywords: newly diagnosed Glioblastoma (WHO Grade IV); Cilengitide; Temozolomide; Radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Cilengitide; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilengitide + Temozolomide + Radiotherapy (Experimental)
  Interventions: Drug: Cilengitide; Drug: Temozolomide; Radiation: Radiotherapy
- Temozolomide + Radiotherapy (Active Comparator)
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cilengitide — Cilengitide 2000 milligram (mg) will be administered intravenously twice weekly over 1 hour infusion from Weeks -1 to 77 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. If considered beneficial in the opinion of the Investigator, continuation of cilengitide treatment will be optional in subjects without disease progression and after Week 77 since start of treatment.
  Arms: Cilengitide + Temozolomide + Radiotherapy
Drug: Temozolomide — Temozolomide (TMZ) 75 milligram per square meter [mg/m^2] will be administered intravenously once daily from Weeks 1 to 6. From Week 11 onwards, TMZ will be given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 or until disease progression.
Radiation: Radiotherapy — Radiotherapy (RTX) at a dose of 2 gray (Gy) per fraction will be given once daily, 5 days per week from Weeks 1 to 6, total dose 60 Gy.

SUMMARY:
CENTRIC is a Phase 3 clinical trial assessing efficacy and safety of the investigational integrin inhibitor, cilengitide, in combination with standard treatment versus standard treatment alone in newly diagnosed glioblastoma subjects with a methylated O6-methylguanine-deoxyribonucleic acid methyltransferase (MGMT) gene promoter in the tumor tissue.

The MGMT gene promoter is a section of deoxyribonucleic acid (DNA) that acts as a controlling element in the expression of MGMT. Methylation of the MGMT gene promoter has been found to be a predictive marker for benefit from temozolomide (TMZ) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor tissue specimens from the glioblastoma surgery or open biopsy (formalin-fixed, paraffin-embedded block; stereotactic biopsy not allowed) must be available for MGMT status analysis and central pathology review
2. Newly diagnosed histologically proven supratentorial glioblastoma (World Health Organization [WHO] Grade IV)
3. Proven methylated MGMT gene promoter methylation status
4. Available post-operative gadolinium-enhanced magnetic resonance imaging (Gd-MRI) performed within less than (<) 48 hours after surgery (in case it was not possible to obtain a Gd-MRI within <48 hours post surgery, a Gd-MRI is to be performed prior to randomization)
5. Stable or decreasing dose of steroids for greater than or equal to (>=) 5 days prior to randomization
6. Eastern Cooperative Oncology Group performance score (ECOG PS) of 0-1
7. Meets 1 of the following recursive partitioning analysis (RPA) classifications: Class III (Age < 50 years and ECOG PS 0). Class IV (meeting one of the following criteria: a) Age < 50 years and ECOG PS 1 or b) Age >= 50 years, underwent prior partial or total tumor resection, mini mental state examination [MMSE] >= 27). Class V (meeting one of the following criteria: a) Age >= 50 years and underwent prior partial or total tumor resection, MMSE < 27 or b) Age >= 50 years and underwent prior tumor biopsy only)
8. Other protocol defined inclusion criteria could apply

Exclusion Criteria:

1. Prior chemotherapy within the last 5 years
2. Prior RTX of the head
3. Receiving concurrent investigational agents or has received an investigational agent within the past 30 days prior to the first dose of cilengitide
4. Prior systemic antiangiogenic therapy
5. Placement of Gliadel® wafer at surgery
6. Inability to undergo Gd-MRI.
7. Planned surgery for other diseases
8. History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months of enrollment
9. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for >= 5 years are eligible for this study
10. History of coagulation disorder associated with bleeding or recurrent thrombotic events
11. Clinically manifest myocardial insufficiency (New York Heart Association [NYHA] III, IV) or history of myocardial infarction during the past 6 months; uncontrolled arterial hypertension
12. Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2008-09; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, Prof. Dr., Study Chair — University of Lausanne Medical Center (CHUV); Andriy Markivskyy, MD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States
- Please Contact the Merck KGaA Communication Center Located in, Darmstadt, Germany

REFERENCES:
- [Result] Cilengitide combined with standard treatment for patients with newly diagnosed glioblastoma with methylated MGMT promoter (CENTRIC EORTC 26071-22072 study): a multicentre, randomised, open-label, phase 3 trial Roger Stupp, Monika E Hegi, Thierry Gorlia, Sara C Erridge, James Perry, Yong-Kil Hong, Kenneth D Aldape, Benoit Lhermitte, Torsten Pietsch, Danica Grujicic, Joachim Peter Steinbach, Wolfgang Wick, Rafał Tarnawski, Do-Hyun Nam, Peter Hau, Astrid Weyerbrock, Martin J B Taphoorn, Chiung-Chyi Shen, Nalini Rao, László Thurzo, Ulrich Herrlinger, Tejpal Gupta, Rolf-Dieter Kortmann, Krystyna Adamska, Catherine McBain, Alba A Brandes, Joerg Christian Tonn, Oliver Schnell, Thomas Wiegel, Chae-Yong Kim, Louis Burt Nabors, David A Reardon, Martin J van den Bent, Christine Hicking, Andriy Markivskyy, Martin Picard, Michael Weller The Lancet Oncology 20 August 2014(Article in Press DOI: 10.1016/S1470-2045(14)70379-1)
- [Derived] Seliger C, Oppong FB, Lefranc F, Chinot O, Stupp R, Nabors B, Gorlia T, Weller M; EORTC Brain Tumor Group. Association of antidepressant drug use with outcome of patients with glioblastoma. Int J Cancer. 2023 Apr 1;152(7):1348-1359. doi: 10.1002/ijc.34344. Epub 2022 Nov 17. PMID 36346112
- [Derived] Stupp R, Hegi ME, Gorlia T, Erridge SC, Perry J, Hong YK, Aldape KD, Lhermitte B, Pietsch T, Grujicic D, Steinbach JP, Wick W, Tarnawski R, Nam DH, Hau P, Weyerbrock A, Taphoorn MJ, Shen CC, Rao N, Thurzo L, Herrlinger U, Gupta T, Kortmann RD, Adamska K, McBain C, Brandes AA, Tonn JC, Schnell O, Wiegel T, Kim CY, Nabors LB, Reardon DA, van den Bent MJ, Hicking C, Markivskyy A, Picard M, Weller M; European Organisation for Research and Treatment of Cancer (EORTC); Canadian Brain Tumor Consortium; CENTRIC study team. Cilengitide combined with standard treatment for patients with newly diagnosed glioblastoma with methylated MGMT promoter (CENTRIC EORTC 26071-22072 study): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1100-8. doi: 10.1016/S1470-2045(14)70379-1. Epub 2014 Aug 19. PMID 25163906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): Sep 2008/Aug 2011. Clinical data cut-off: 19 Nov 2012, Study completion date: Aug 2013.
Pre-assignment Details: Enrolled: 3471 screened for eligibility; 2926 excluded (mainly due to unmethylated O6-methylguanine-DNA methyltransferase status and non-fulfillment of inclusion or exclusion criteria), 545 participants randomized.
Groups:
- Cilengitide + Temozolomide + Radiotherapy: Cilengitide 2000 milligram (mg) twice weekly over 1 hour intravenous infusion from Weeks -1 to 77, Temozolomide (TMZ) 75 milligram per square meter [mg/m^2] intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and radiotherapy (RTX) at a dose of 2 Gray (Gy) per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. Continuation of cilengitide treatment after Week 77 was optional in participants without disease progression, If considered beneficial in the opinion of the Investigator.
- Temozolomide + Radiotherapy: TMZ 75 mg/m^2 administered intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and RTX at a dose of 2 Gy per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason.
Period: Overall Study
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Started | 272 | 273
Completed | 233 | 237
Not Completed | 39 | 36
Not completed — Ongoing at cut-off date | 39 | 36

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy | Total
Number analyzed (Participants) | 272 | 273 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.00) | 56.0 (10.97) | 56.4 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 130 | 254
  Male | 148 | 143 | 291

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: The OS time is defined as the time (in months) from randomization to death or last day known to be alive. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, that is, Sep 2008 until cut-off date, (19 Nov 2012)
Population: ITT population included all the participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 272 | 273
Months | 26.3 [23.8 to 28.8] | 26.3 [23.9 to 34.7]
Statistical Analysis 1: Comparison: Cilengitide + Temozolomide + Radiotherapy vs Temozolomide + Radiotherapy; Test type: Superiority or Other; p = 0.8623, Log Rank — P-value is not adjusted for multiple testing; Hazard Ratio (HR) = 1.021, 95% CI 2-sided [0.808 to 1.291]

2. Secondary Outcome: Progression Free Survival (PFS) Time - Investigator and Independent Read
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause. Investigator read is the assessment of all imaging by the treating physician at the local trial site and Independent Read is the assessment of all imaging centrally by an Independent Review Committee (IRC). Investigator's assessed progression according to MacDonald criteria and IRC by Response Assessment in Neuro-Oncology Working Group (RANO) criteria using Gadolinium-enhanced magnetic resonance imaging.
  Investigator and IRC read: Progression is defined as greater than 25 percent increase in the sum of the product of the largest perpendicular diameters of enhancing tumor compared to the smallest prior sum, or Worsening of an evaluable lesion(s),or Marked increase in T2/FLAIR non-enhancing lesions (IRC only) or Any new lesion
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, Sep 2008 until cut-off date, (19 Nov 2012)
Population: ITT population included all the participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 272 | 273
Months
  PFS Time: Investigator read | 13.5 [10.8 to 15.9] | 10.7 [8.1 to 13.3]
  PFS Time: Independent read | 10.6 [8.2 to 13.4] | 7.9 [5.9 to 12.5]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2.1.
Time Frame: Day 1 of Week -1
Population: Analysis population included all participants of "Cilengitide + Temozolomide + Radiotherapy" group who received at least 1 cilengitide dose with plasma concentration data available on Day 1 of Week -1.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cilengitide + Temozolomide + Radiotherapy
Number analyzed (Participants) | 38
nanogram per milliliter (ng/mL) | 167363.2 (368301.11)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: The Tmax for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2.1.
Time Frame: Day 1 of Week -1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cilengitide + Temozolomide + Radiotherapy
Number analyzed (Participants) | 38
hours | 1.029 (0.401)

5. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to 6 Hours (AUC [0-6]) After Dose
Description: The AUC (0-6) for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2.1.
Time Frame: Day 1 of Week -1
Population: Analysis population included all participants of "Cilengitide + Temozolomide + Radiotherapy" group who received at least 1 cilengitide dose with plasma concentration data available on Day 1 of Week -1. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Cilengitide + Temozolomide + Radiotherapy
Number analyzed (Participants) | 37
hour*ng/mL | 295171.2 (198050.62)

6. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Sub-scale Scores
Description: The EORTC QLQ-C30 is a questionnaire including following sub-scales: global health status, functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social activity), symptom scales (fatigue, nausea and vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties). Scores are averaged for each scale and transformed to 0-100 scale; higher score indicates better quality of life on global health status and functional scales and worse quality of life on symptom scales and financial difficulty scale.
Time Frame: Up to 50 months
Population: ITT population included all the participants who were randomized to study treatment. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 71 | 93
units on a scale
  Global Health Status (n=71, 92) | 54.34 (25.58) | 55.43 (27.02)
  Physical Functioning (n=71, 92) | 65.70 (33.01) | 67.46 (31.19)
  Role Functioning (n=71, 92) | 56.34 (37.31) | 56.34 (35.19)
  Emotional Functioning (n=71, 93) | 67.49 (30.58) | 67.00 (27.29)
  Cognitive Functioning (n=70, 93) | 64.05 (29.16) | 65.41 (31.40)
  Social Activity (n=71, 93) | 56.34 (36.77) | 62.72 (35.73)
  Fatigue (n=71, 92) | 44.37 (33.07) | 39.73 (29.93)
  Nausea and Vomiting (n=71, 93) | 10.33 (20.77) | 7.71 (16.03)
  Pain (n=71, 93) | 22.30 (29.40) | 24.37 (28.93)
  Dyspnoea (n=71, 92) | 15.96 (28.09) | 13.04 (22.62)
  Insomnia (n=71, 91) | 20.66 (30.01) | 20.51 (26.65)
  Appetite Loss (n=71, 92) | 21.13 (30.47) | 15.94 (28.59)
  Constipation (n=71, 93) | 18.78 (28.02) | 13.98 (25.69)
  Diarrhoea (n=70, 92) | 6.67 (18.48) | 4.35 (13.28)
  Financial Difficulties (n=71, 93) | 27.23 (31.53) | 22.94 (31.46)

7. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Brain Module (EORTC QLQ-BN20) Sub-scale Scores
Description: The QLQ-BN20 is a questionnaire specifically designed as the QLQ-C30 supplement for the evaluation of quality of life in brain tumor participants. It includes 4 multi-item sub-scales: future uncertainty, visual disorder, motor dysfunction, communication deficits, and 7 single-item scales: headaches, seizures, drowsiness, itchy skin, hair loss, weakness of legs, and bladder control. All items are rated on a 4-point Likert-type scale ('1=not at all', '2=a little', '3=quite a bit' and '4=very much'), and are linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Time Frame: Up to 50 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 68 | 87
units on a scale
  Future Uncertainty (n=68, 86) | 44.49 (29.70) | 39.31 (30.24)
  Visual Disorder (n=68, 85) | 12.99 (20.24) | 17.78 (23.77)
  Motor Dysfunction (n=68, 86) | 27.45 (30.62) | 23.39 (25.95)
  Communication Deficit (n=68, 86) | 26.14 (28.59) | 19.96 (27.89)
  Headaches (n=68, 86) | 25.98 (32.50) | 21.71 (26.45)
  Seizures (n=68, 87) | 9.31 (22.93) | 8.05 (20.94)
  Drowsiness (n=66, 87) | 38.38 (33.71) | 35.25 (31.07)
  Itchy Skin (n=68, 86) | 9.80 (20.00) | 13.57 (24.72)
  Hair Loss (n=66, 86) | 13.13 (22.55) | 15.12 (26.40)
  Weakness of Legs (n=67, 85) | 24.38 (34.12) | 20.39 (28.68)
  Bladder Control (n=67, 85) | 19.40 (29.67) | 10.20 (21.22)

8. Secondary Outcome: EuroQol 5-Dimensions (EQ-5D) Questionnaire Index
Description: The EuroQuol-5D (EQ-5D) questionnaire is a measure of health status that provides a simple descriptive profile and a single index value. The optional part of the questionnaire was not applied. The EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 5 items are combined to generate health profiles. These profiles were converted to a continuous single index score using a one to one matching. The lowest possible score is -0.594 (death) and the highest is 1.00 (full health).
Time Frame: Up to 50 months
Population: ITT population included all the participants who were randomized to study treatment. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 69 | 90
units on a scale | 0.598 (0.43) | 0.623 (0.36)

9. Secondary Outcome: Number of Participants With Change From Baseline in Work Status at End of Study
Description: Number of participants with change from baseline in work status (working full time [FT], part-time [PT], unemployed/retired [U/R]) at end of study (EOS) (up to cut-off date, [19 Nov 2012]) was reported. For the category 'part-time', the following sub-categories were defined: part-time due to basic disease (PT1); part-time not due to basic disease (PT2); part-time reason not known (PT3).
Time Frame: Baseline, End of study (up to cut-off date, [19 Nov 2012])
Population: Safety population included all the participants who received any dose of study treatment that is Cilengitide, Temozolomide or Radiotherapy. According to trial design safety data in trial arms (Cilengitide vs Control) were collected based on different visit frequency and different safety surveillance period.
Measure: Number; unit: participants
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 263 | 258
participants
  Baseline: FT, EOS: FT | 3 | 6
  Baseline: FT, EOS: PT1 | 2 | 1
  Baseline: FT, EOS: PT2 | 1 | 0
  Baseline: FT, EOS: PT3 | 0 | 0
  Baseline: FT, EOS: U/R | 24 | 22
  Baseline: PT1, EOS: FT | 3 | 2
  Baseline: PT1, EOS: PT1 | 3 | 1
  Baseline: PT1, EOS: PT2 | 0 | 0
  Baseline: PT1, EOS: PT3 | 0 | 0
  Baseline: PT1, EOS: U/R | 9 | 12
  Baseline: PT2, EOS: FT | 0 | 1
  Baseline: PT2, EOS: PT1 | 0 | 0
  Baseline: PT2, EOS: PT2 | 0 | 0
  Baseline: PT2, EOS: PT3 | 1 | 0
  Baseline: PT2, EOS: U/R | 5 | 4
  Baseline: PT3, EOS: FT | 0 | 0
  Baseline: PT3, EOS: PT1 | 0 | 0
  Baseline: PT3, EOS: PT2 | 0 | 0
  Baseline: PT3, EOS: PT3 | 0 | 0
  Baseline: PT3, EOS: U/R | 0 | 0
  Baseline: U/R, EOS: FT | 5 | 8
  Baseline: U/R, EOS: PT1 | 5 | 7
  Baseline: U/R, EOS: PT2 | 1 | 1
  Baseline: U/R, EOS: PT3 | 0 | 0
  Baseline: U/R, EOS: U/R | 199 | 191
  Baseline: Missing, EOS: FT | 0 | 0
  Baseline: Missing, EOS: PT1 | 0 | 0
  Baseline: Missing, EOS: PT2 | 0 | 0
  Baseline: Missing, EOS: PT3 | 0 | 0
  Baseline: Missing, EOS: U/R | 1 | 1
  Baseline: Missing, EOS: Missing | 1 | 1

10. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, Treatment-Related AEs, Treatment-Related Serious AEs, AEs Leading to Death, Treatment Related AEs Leading to Death, AEs of Grade 3 or 4 and Treatment Related AEs of Grade 3 or 4
Description: An AE is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. Treatment-emergent AEs are the events between first dose of study drug and up to 28 days after last dose of study treatment. A Serious AE is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-related AEs are the AEs which are suspected to be reasonably related to the study treatment (cilengitide, or radiotherapy, or temozolomide) as per investigator assessment. The severity of AEs was assessed according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTCAE) (version 3.0): Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling. Note: Death (Grade 5) was regarded as an outcome.
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first participant randomized, that is, Sep 2008 until cut-off date (19 Nov 2012)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 263 | 258
Participants
  AEs | 261 | 253
  Serious AEs | 138 | 115
  Treatment-related AEs | 229 | 222
  Treatment-Related Serious AEs | 55 | 47
  AEs leading to death | 11 | 9
  Treatment-related AEs leading to death | 3 | 3
  AEs with NCI-CTC toxicity Grade 3 or 4 | 169 | 158
  Treatment-related AEs of Grade 3 or 4 | 100 | 101

11. Secondary Outcome: Number of Participants With AEs Belonging to Standardized Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs) Thromboembolic Events and Hemorrhage With NCI-CTC Toxicity Grade 3 or 4
Description: Thromboembolic events (standardized MedDRA query [SMQ]) Grade 3 or 4 AEs encompassed hemiparesis and cerebrovascular accident, pulmonary embolism, and deep vein thrombosis. Thromboembolic events (SMQ) of any grade and of Grade 3 or 4 were generally more frequent in the Cilengitide + Temozolomide/Radiotherapy group than in the Temozolomide/Radiotherapy group but were still in the expected range of this patient population The severity of AEs was assessed according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTCAE) (version 3.0): Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling. Note: Death (Grade 5) was regarded as an outcome.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 263 | 258
Participants
  SMQ:Thromboembolic events | 35 | 23
  SMQ: Hemorrhage | 4 | 4

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) and Lab Parameters
Time Frame: Up to 50 months
Population: Any clinically significant abnormal ECG and lab finding was planned to be reported as AE only so they have been captured in the below mentioned adverse event section.
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first participant randomized, that is, Sep 2008 until cut-off date (19 Nov 2012)
Groups:
- Cilengitide + Temozolomide + Radiotherapy: Cilengitide 2000 milligram (mg) twice weekly over 1 hour intravenous infusion from Weeks -1 to 77, Temozolomide (TMZ) 75 milligram per square meter [mg/m^2] intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and radiotherapy (RTX) at a dose of 2 gray (Gy) per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. Continuation of cilengitide treatment after Week 77 will be optional in participants without disease progression, If cilengitide treatment considered beneficial in the opinion of the Investigator,
Arm/Group | Cilengitide + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Serious Adverse Events (participants affected / at risk) | 138/263 | 115/258
Other Adverse Events (participants affected / at risk) | 251/263 | 240/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide + Temozolomide + Radiotherapy (N=263) | Temozolomide + Radiotherapy (N=258)
CONVULSION (Nervous system disorders) | 20 | 14
HEMIPARESIS (Nervous system disorders) | 12 | 1
BRAIN OEDEMA (Nervous system disorders) | 5 | 5
EPILEPSY (Nervous system disorders) | 6 | 3
GRAND MAL CONVULSION (Nervous system disorders) | 5 | 3
HEADACHE (Nervous system disorders) | 5 | 1
PARTIAL SEIZURES (Nervous system disorders) | 4 | 2
STATUS EPILEPTICUS (Nervous system disorders) | 4 | 1
COGNITIVE DISORDER (Nervous system disorders) | 3 | 1
DIZZINESS (Nervous system disorders) | 3 | 1
SOMNOLENCE (Nervous system disorders) | 3 | 1
ATAXIA (Nervous system disorders) | 2 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 | 0
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 2 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 | 0
APHASIA (Nervous system disorders) | 1 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 1
SPEECH DISORDER (Nervous system disorders) | 2 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 0
BRAIN INJURY (Nervous system disorders) | 1 | 0
CENTRAL NERVOUS SYSTEM NECROSIS (Nervous system disorders) | 1 | 0
CEREBRAL CYST (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 | 1
COMA (Nervous system disorders) | 0 | 1
COORDINATION ABNORMAL (Nervous system disorders) | 1 | 0
FACIAL NERVE DISORDER (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 1 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 0 | 1
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 1 | 0
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 | 1
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 | 0
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 | 0
VISUAL FIELD DEFECT (Nervous system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 | 24
NEUTROPENIA (Blood and lymphatic system disorders) | 6 | 11
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 10
ANAEMIA (Blood and lymphatic system disorders) | 2 | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
HAEMATOTOXICITY (Blood and lymphatic system disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 9 | 7
URINARY TRACT INFECTION (Infections and infestations) | 2 | 4
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0
CELLULITIS (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 1
H1N1 INFLUENZA (Infections and infestations) | 1 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 1
SEPSIS (Infections and infestations) | 2 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 2
WOUND INFECTION (Infections and infestations) | 2 | 0
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1
WOUND ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BRAIN ABSCESS (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 1 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 1
MENINGITIS (Infections and infestations) | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 12 | 7
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 4 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PYREXIA (General disorders) | 4 | 3
ASTHENIA (General disorders) | 5 | 1
FATIGUE (General disorders) | 4 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 3
DISEASE PROGRESSION (General disorders) | 4 | 0
DEVICE MALFUNCTION (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
GAIT DISTURBANCE (General disorders) | 1 | 0
PAIN (General disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 3 | 4
NAUSEA (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 1
ENTERITIS (Gastrointestinal disorders) | 2 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRIC DISORDER (Gastrointestinal disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 5 | 6
HYPOTENSION (Vascular disorders) | 3 | 1
HYPERTENSION (Vascular disorders) | 1 | 2
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 1 | 1
THROMBOSIS (Vascular disorders) | 0 | 1
EMBOLISM VENOUS (Vascular disorders) | 1 | 0
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 5 | 2
AGITATION (Psychiatric disorders) | 0 | 3
DEPRESSION (Psychiatric disorders) | 1 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
DISORIENTATION (Psychiatric disorders) | 1 | 0
DYSTHYMIC DISORDER (Psychiatric disorders) | 1 | 0
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
PANIC ATTACK (Psychiatric disorders) | 0 | 1
PERSONALITY CHANGE (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1
SCHIZOPHRENIA (Psychiatric disorders) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 2
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 1
OPEN WOUND (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL OEDEMA (Injury, poisoning and procedural complications) | 0 | 1
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
RADIATION INJURY (Injury, poisoning and procedural complications) | 0 | 1
RADIATION NECROSIS (Injury, poisoning and procedural complications) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 | 1
PLATELET COUNT DECREASED (Investigations) | 2 | 1
BLOOD URIC ACID INCREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
FIBRIN D DIMER INCREASED (Investigations) | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 0
TRANSAMINASES INCREASED (Investigations) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTRACRANIAL TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEURILEMMOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CORONARY ARTERY THROMBOSIS (Cardiac disorders) | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 1
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 1 | 0
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
BLADDER CATHETERISATION (Surgical and medical procedures) | 1 | 0
PALLIATIVE CARE (Surgical and medical procedures) | 0 | 1
SURGERY (Surgical and medical procedures) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 1
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 | 1
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide + Temozolomide + Radiotherapy (N=263) | Temozolomide + Radiotherapy (N=258)
NAUSEA (Gastrointestinal disorders) | 128 | 125
CONSTIPATION (Gastrointestinal disorders) | 100 | 78
VOMITING (Gastrointestinal disorders) | 77 | 83
DIARRHOEA (Gastrointestinal disorders) | 44 | 20
DYSPEPSIA (Gastrointestinal disorders) | 24 | 8
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 6
HEADACHE (Nervous system disorders) | 114 | 87
DIZZINESS (Nervous system disorders) | 33 | 24
CONVULSION (Nervous system disorders) | 37 | 14
MEMORY IMPAIRMENT (Nervous system disorders) | 27 | 17
APHASIA (Nervous system disorders) | 24 | 11
TREMOR (Nervous system disorders) | 20 | 11
PARAESTHESIA (Nervous system disorders) | 14 | 7
FATIGUE (General disorders) | 98 | 84
ASTHENIA (General disorders) | 42 | 20
OEDEMA PERIPHERAL (General disorders) | 36 | 24
PYREXIA (General disorders) | 26 | 16
ALOPECIA (Skin and subcutaneous tissue disorders) | 70 | 70
PRURITUS (Skin and subcutaneous tissue disorders) | 32 | 15
RASH (Skin and subcutaneous tissue disorders) | 28 | 18
ERYTHEMA (Skin and subcutaneous tissue disorders) | 21 | 10
DRY SKIN (Skin and subcutaneous tissue disorders) | 16 | 12
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 46 | 46
LYMPHOPENIA (Blood and lymphatic system disorders) | 45 | 35
LEUKOPENIA (Blood and lymphatic system disorders) | 29 | 23
NEUTROPENIA (Blood and lymphatic system disorders) | 29 | 18
ANAEMIA (Blood and lymphatic system disorders) | 15 | 15
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 28 | 16
NASOPHARYNGITIS (Infections and infestations) | 32 | 11
URINARY TRACT INFECTION (Infections and infestations) | 16 | 21
DECREASED APPETITE (Metabolism and nutrition disorders) | 53 | 45
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 31 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 24 | 13
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 21 | 14
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 25 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 51 | 23
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 8
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 20 | 6
INSOMNIA (Psychiatric disorders) | 35 | 24
DEPRESSION (Psychiatric disorders) | 19 | 14
ANXIETY (Psychiatric disorders) | 13 | 14
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 21 | 17
WEIGHT DECREASED (Investigations) | 15 | 14
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 20 | 22
VISION BLURRED (Eye disorders) | 16 | 11
HYPERTENSION (Vascular disorders) | 17 | 7
URINARY INCONTINENCE (Renal and urinary disorders) | 15 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All manuscripts and materials relating to Study shall be submitted to Sponsor at least 60 days prior to submitting/presenting and allow Sponsor 60 days for review. If Sponsor requests, any confidential information shall be removed. In multi-center study, any publication shall not be made before the first multi-center publication; provided, however, that if no multi-center publication is made within 1 year from database lock, then Site may publish individually in accordance with this provision.